CLINICAL TRIAL: NCT06139640
Title: The Effect of Damask Rose Essential Oil Aromatherapy on Dental Anxiety and Pain on Children Undergoing Local Anesthesia: A Randomized Clinical Trial
Brief Title: The Effect of Damask Rose Essential Oil Aromatherapy on Dental Anxiety and Pain on Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Moushtaha Sayed Hamid (Other)
Collaborators: clinical professor (Unknown)
Responsible Party: Sponsor-Investigator, Moushtaha Sayed Hamid, principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: Aromatherapy on Dental Anxiety
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-11

CONDITIONS: Dental Anxiety
Keywords: Aromatherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The effects of rose oil on pain and anxiety level on pediatric dental patient (Active Comparator): Rose oil aromatherapy
  Interventions: Other: Damask Rose Essential Oil
- The effects of no treatment on pain and anxiety level on pediatric dental patient (No Intervention)

INTERVENTIONS:
Other: Damask Rose Essential Oil — Aromatherapy is a relaxation therapy media that uses aromatic essence extracts from plant parts. Aromatherapy is used to treat and improve physical and psychological health
  Arms: The effects of rose oil on pain and anxiety level on pediatric dental patient

SUMMARY:
This study aims to Evaluate and compare the role of Damask rose essential oils in reducing a child's dental anxiety and pain undergoing local anesthesia administration

DETAILED DESCRIPTION:
Dental anxiety is recognized as one of the major public health problems. It can lead to avoidance of necessary dental care, which affects oral health negatively, especially in children where dental care providers face a challenge to control dental anxiety to manage the child in the dental visit. Overall prevalence of dental anxiety was 23.9% with less prevalent in adolescents (13.3%), more prevalent in preschoolers (36.5%), and schoolchildren (25.8%).

Methods for managing anxiety in dentistry are both pharmacological and non-pharmacological. Aromatherapy is one of the non-pharmacological methods, it is a Simple, inexpensive, non-invasive method introduced by the use of aromatic essential oils through the sense of smell to produce positive physiological effects, relaxation and relieve anxiety symptoms. Aromatherapy can also decrease pain perception during local anesthetic injections in children.

Rosa damascene is commonly known as Damask roses, a plant belonging to the Rosaceae family. The flowers of this plant are large, showy and colorful. for its scent, it is also used in the production of essential oil and rose water. The R. damascena plant has also been used for medicinal applications it has analgesic, anti-inflammatory, anti-headache, and muscle-relaxing effects, and due to its strong depressing effect on the central nervous system it has hypnotic, anticonvulsant, antidepressant, and ant anxiety, effects.

The effect of rose oil in reducing pain has been conducted in children who are hospitalized for surgery, measuring the effect on post-operative pain intensity. Also, the effect of rose oil in the reduction of dental anxiety has already been studied but has been conducted on adults orthodontic patients.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian children from 7 to 12 years old require local anesthesia administration.
* Absence of any systemic problems, physical and mental disabilities.
* Children intellectually sufficient to complete the anxiety scale and those whose parents were willing to participate in the study.
* Frankel rating 3 in cooperation

Exclusion Criteria:

* Presence of dental or medical emergency and systemic disorders.
* Special needs children.
* Children with any respiratory tract illnesses, common, cold or allergy.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pulse rate | immediately after the intervention
  will be recorded by an Automated blood pressure device

SECONDARY OUTCOMES:
Level of anxiety | immediately after the intervention
  will be recorded by Dental Anxiety Scale - Faces version [16] Modified Child Dental Anxiety Scale simplified Scores (1-5) higher scores mean worse outcome
Blood pressure (systolic and diastolic blood pressure) | immediately after the intervention
  will be recorded by an Automated blood pressure device
Pain rating scale | immediately after the intervention
  will be recorded by Faces, legs, activity, cry, and controllability scale (FLACC) Score(0-10) higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kamal El-Motayam, Professor, Study Director — Professor

IPD SHARING:
Plan to Share IPD: No